CLINICAL TRIAL: NCT05428111
Title: Expression of Programmed Death-1 (PD-1) & Programmed Death Ligand-1 (PDL-1) in Acute Lymphoblastic Leukemia in Pediatric
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nada Mohamed Rafat, resident doctor at clinical pathology department at sohag oncology center, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-22-06-10
Record Dates: First submitted 2022-06-15; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Acute Lymphoblastic Leukemia in Pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): healthy control individuals
  Interventions: Diagnostic Test: flow cytometric immunophynotyping
- case (Active Comparator): Newly diagnosed and under treatment cases of acute lymphoblastic leukemic
  Interventions: Diagnostic Test: flow cytometric immunophynotyping

INTERVENTIONS:
Diagnostic Test: flow cytometric immunophynotyping — Expression of programmed death-1 (PD-1) & programmed death ligand-1 (PDL-1) in flow cytometric immunophynotyping

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common childhood malignancy in the world.

It is a malignant clonal proliferation of lymphoid progenitor cells, but most commonly of the B cell lineage (B ALL). .

Acute Lymphoblastic Leukemia (ALL) is a heterogeneous disease that causes malignant hematological disorders at any age. It mainly affects children aged 2 to 5; in fact, 60% of pediatric leukemia cases are ALL, with an incidence of 3-4 cases per 100,000 per year. It is divided into two subtypes B-ALL and T-ALL depending on whether transformation occurs in B- or T-cell precursors, respectively .

Leukemic cells apply multiple immune evasion mechanisms resulting in tumor progression. One of the most important immune escape mechanisms is over expression of immune checkpoint receptors and their ligands such as PD-1 and PD-L1 .

The PD-1 receptor plays a crucial role in a broad spectrum of immune regulatory mechanisms .

It is a negative co-receptor that down regulates T-cell activity .

PDL 1, which is known as B7 H1 , is a cell surface protein of B7 family member .

PD L1 is expressed on all types of lympho hematopoietic cells at variable levels and is constitutively expressed on T cells, B cells, macrophages, and dendritic cells .

Tumors exploit the PD-1/PD-L1 pathway to evade host immune surveillance .

PD-1/PD-L1 pathway controls the induction and maintenance of immune tolerance within the tumor microenvironment. The activity of PD-1 and its ligands PD-L1 or PD-L2 are responsible for T cell activation, proliferation, and cytotoxic secretion in cancer to produce anti-tumor immune responses .

ELIGIBILITY:
Inclusion Criteria:

* Age range from 1 day to 18 years old
* Patients who are newly diagnosed and under treatment of acute lymphoblastic leukemia

Exclusion Criteria:

* Other types of acute leukemia rather than acute lymphoblastic leukemia

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
programmed death-1 (PD-1) by flow cytometry immunophynotyping | 6 months
  Assess programmed death-1 by flow cytometry immunophynotyping
Programmed death ligand -1 (PDL-1) by flow cytometry immunophynotyping | 6 months
  Assess programmed death ligand -1 by flow cytometry immunophynotyping

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Taghiloo S, Asgarian-Omran H. Immune evasion mechanisms in acute myeloid leukemia: A focus on immune checkpoint pathways. Crit Rev Oncol Hematol. 2021 Jan;157:103164. doi: 10.1016/j.critrevonc.2020.103164. Epub 2020 Nov 18. PMID 33271388
- [Background] Bergman PJ, Clifford CA. Recent Advancements in Veterinary Oncology. Vet Clin North Am Small Anim Pract. 2019 Sep;49(5):xiii-xiv. doi: 10.1016/j.cvsm.2019.06.001. No abstract available. PMID 31345517
- [Background] Woo JS, Alberti MO, Tirado CA. Childhood B-acute lymphoblastic leukemia: a genetic update. Exp Hematol Oncol. 2014 Jun 13;3:16. doi: 10.1186/2162-3619-3-16. eCollection 2014. PMID 24949228
- [Background] Chiaretti S, Vitale A, Cazzaniga G, Orlando SM, Silvestri D, Fazi P, Valsecchi MG, Elia L, Testi AM, Mancini F, Conter V, te Kronnie G, Ferrara F, Di Raimondo F, Tedeschi A, Fioritoni G, Fabbiano F, Meloni G, Specchia G, Pizzolo G, Mandelli F, Guarini A, Basso G, Biondi A, Foa R. Clinico-biological features of 5202 patients with acute lymphoblastic leukemia enrolled in the Italian AIEOP and GIMEMA protocols and stratified in age cohorts. Haematologica. 2013 Nov;98(11):1702-10. doi: 10.3324/haematol.2012.080432. Epub 2013 May 28. PMID 23716539
- [Derived] Allam AA, Ahmed HA, Hassan MA, Khaled SAA, Shibl A, Osman AM, Ali NMR, Ahmed NM. Programmed Cell Death-1 and Programmed Cell Death Ligand-1 in Childhood Acute B-Lymphoblastic Leukemia: Expression and Significance as Biomarker. Int J Lab Hematol. 2025 Oct;47(5):832-839. doi: 10.1111/ijlh.14472. Epub 2025 Apr 1. PMID 40166836